CLINICAL TRIAL: NCT03193528
Title: A Novel Multiplex ELISA Assay for Evaluating Patients With Gross Hematuria for Bladder Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); University of Texas (Other); Nara Medical University (Other); University of California, Los Angeles (Other); Nonagen Bioscience Corporation (Industry); National Cancer Institute (NCI) (NIH); University of Rochester (Other); Nara Prefecture Seiwa Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: Rosser-2015-7; R01CA198887 (NIH)
Record Dates: First submitted 2017-06-17; First posted 2017-06-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine collection (minimal 50 mL) and cystoscopy (+ biopsy w/in 4 weeks, if abnormal noted)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To improve upon the non-invasive detection of BCa by further validating a multiplex ELISA assay directed at a BCa-associated diagnostic signature in voided urine samples of patients with gross hematuria.

DETAILED DESCRIPTION:
Hematuria is the most common presentation of BCa with 22% of patients with gross hematuria harboring BCa. VUC is the most widely used urine-based assay for detecting BCa; however, it fails to detect approximately 50% of low-grade or early stage BCa when it is most curable.

Because of this severe limitation, patients with hematuria (microscopic or gross) will undergo an invasive examination of the urinary bladder, where a miniature camera is inserted into the bladder. We propose to improve upon the non-invasive detection of BCa by further validating a multiplex ELISA assay directed at a BCa-associated diagnostic signature in voided urine samples of patients with gross hematuria.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have documented or reported gross hematuria within 3 month of study enrollment
* Willing and able to give written informed consent

Exclusion Criteria (patients must not):

* Have history of BCa
* History of previous cancer (excluding basal and squamous cell skin cancer) within the past 3 years
* Have a known active urinary tract infection or urinary retention
* Have active stone disease (renal or bladder) or renal insufficiency (creatinine >2.0 mg/dL) Serum creatinine value can be up to 60 days before consent, otherwise repeat
* Have ureteral stents, nephrostomy tubes or bowel interposition
* Have recent genitourinary instrumentation (within 10 days prior to signing consent)
* Be unable or unwilling to complete the hematuria evaluation (i.e., cystoscopy and upper tract imaging)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, age 18 and older who have documented gross hematuria within the past 3 months who are referred for cystoscopy and are willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To examine the sensitivity and specificity of the multiplex ELISA assay directed at a BCa-associated diagnostic signature in voided urine samples to reference standard of cystoscopy in a cohort of 450 participants presenting with gross hematuria. | 1 year

SECONDARY OUTCOMES:
To compare the sensitivity and specificity of the multiplex ELISA assay to VUC and NMP22® BladderChek to reference standard of cystoscopy in this cohort. | 1 year
To develop a BCa risk calculator from this cohort using cutting edge machine learning techniques (e.g., random forest) incorporating biomarker data and clinical data. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rosser, MD, Study Director — Nonagen Bioscience Corporation; Hideki Furuya, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (6):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of Rochester Medical Center, Rochester, New York
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
- Japan (2):
  - Department of Urology, Nara Medical University, Nara
  - Nara Precfecture Seiwa Medical Center, Nara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. J Transl Med. 2024 Jan 2;22(1):8. doi: 10.1186/s12967-023-04811-2. PMID 38167321
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. Res Sq [Preprint]. 2023 Nov 25:rs.3.rs-3635581. doi: 10.21203/rs.3.rs-3635581/v1. PMID 38045238

DOCUMENTS (1):
  • Informed Consent Form (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT03193528/ICF_000.pdf